CLINICAL TRIAL: NCT02243280
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Co-Administration of ABT-493 and ABT-530 With and Without Ribavirin in Subjects With Chronic Hepatitis C Virus (HCV) Genotype 1, 4, 5, and 6 Infection (SURVEYOR-I)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Co-administration of ABT-493 and ABT-530 With and Without Ribavirin in Subjects With HCV Genotype 1, 4, 5, and 6 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-867; 2014-002925-36 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-09-17 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus; HCV
Keywords: HCV GT4; Hepatitis C virus; HCV GT1; HCV; Compensated Cirrhosis; HCV GT6; Hepatitis C Genotype 4 (GT 4); Hepatitis C Genotype 1 (GT1); RBV; Cirrhotic; Hepatitis C; Interferon (IFN) Free; IFN free; HCV GT5; Chronic Hepatitis C; Ribavirin; Child Pugh A; Hepatitis C Genotype 5 (GT 5); Hepatitis C Genotype 6 (GT 6); ABT-493; ABT-530; glecaprevir; pibrentasvir
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Arm A (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 120 mg QD for 12 weeks in HCV genotype 1-infected participants without cirrhosis
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm B (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 40 mg QD for 12 weeks in HCV genotype 1- infected participants without cirrhosis
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm C (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 120 mg QD for 8 weeks in HCV genotype 1-infected participants without cirrhosis (never opened - Sponsor decision)
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm D (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 40 mg QD for 8 weeks in HCV genotype 1-infected participants without cirrhosis (never opened - Sponsor decision)
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm E (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 120 mg QD + ribavirin (RBV) 800 mg QD for 12 weeks in HCV genotype 1-infected participants with compensated cirrhosis (never opened - Sponsor decision)
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm F (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 120 mg QD for 12 weeks in HCV genotype 1- infected participants with compensated cirrhosis
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm G (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 40 mg QD + ribavirin (RBV) 800 mg QD for 12 weeks in HCV genotype 1-infected participants with compensated cirrhosis (never opened - Sponsor decision)
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm H (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 40 mg QD for 12 weeks in HCV genotype 1-infected participants with compensated cirrhosis (never opened - Sponsor decision)
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm I (Experimental): ABT-493 300 mg once daily (QD) + ABT-530 120 mg QD for 12 weeks in HCV genotype 4-, 5-, and 6-infected participants without cirrhosis
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm J (Experimental): ABT-493 200 mg once daily (QD) + ABT-530 40 mg QD for 12 weeks in HCV genotype 4-, 5-, and 6-infected participants without cirrhosis (never opened - Sponsor decision)
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm K (Experimental): ABT-493 300 mg once daily (QD) + ABT-530 120 mg QD for 8 weeks in HCV genotype 1- infected participants without cirrhosis
  Interventions: Drug: ABT-493; Drug: ABT-530

INTERVENTIONS:
Drug: ABT-493 — Tablet
  Other Names: glecaprevir
Drug: ABT-530 — Tablet
  Other Names: pibrentasvir

SUMMARY:
The purpose of this Phase 2, open-label, 2-part, multicenter study was to evaluate the efficacy, safety, and pharmacokinetics of co-administration of ABT-493 and ABT-530 with and without ribavirin (RBV) at different doses in chronic Hepatitis C virus (HCV) Genotype 1 (GT1), Genotype 4 (GT4), Genotype 5 (GT5), and Genotype 6 (GT6) infection with compensated cirrhosis (GT1 only) or without cirrhosis (GT1, GT4, GT5, or GT6). Although RBV was initially planned in the protocol, it was not administered in any of the study arms.

DETAILED DESCRIPTION:
This study consisted of two independent parts: Part 1 was conducted first followed by Part 2. Part 1 enrolled participants who received ABT-493 and ABT-530 for 12 weeks; Part 2 enrolled participants who received ABT-493 and ABT-530 for 8 or 12 weeks. Participants who completed or prematurely discontinued the treatment period were followed for 24 weeks to monitor HCV RNA to evaluate efficacy and the emergence and persistence of viral variants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 70 years of age, inclusive, at time of screening
2. Screening laboratory result indicating hepatitis C virus (HCV) GT1 (Study Parts 1 and 2) or GT4, GT5, or GT6 (Study Part 2) infection
3. Chronic HCV infection defined as one of the following:

   * Positive for anti-HCV antibody (Ab) or HCV RNA at least 6 months before screening, and positive for HCV RNA and anti-HCV Ab at the time of screening or
   * Positive for anti-HCV Ab and HCV RNA at the time of screening with a liver biopsy consistent with chronic HCV infection (or a liver biopsy performed prior to enrollment with evidence of chronic HCV infection)
4. Participant had to meet one of the following criteria:

   * Treatment-naïve: participant had never received treatment for HCV infection
   * Treatment-experienced: pegylated-interferon alpha-2a or alpha-2b and ribavirin (PR)-null responder (for Study Part 1) or PR-experienced (on-treatment failure or prior relapse) (for Study Part 2)
5. Documented absence of cirrhosis (in Study Part 1 and in corresponding arms of Study Part 2), or compensated cirrhosis (in corresponding arms of Study Part 2, GT1 only), per local standard

Exclusion Criteria:

1. History of severe, life-threatening or other significant sensitivity to any drug
2. Female who is pregnant, planning to become pregnant during the study or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study
3. Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator
4. Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab)
5. Hepatitis C virus (HCV) genotype performed during screening indicating co-infection with more than one HCV genotype
6. Any cause of liver disease other than chronic HCV infection
7. Participants with plasma HCV RNA load ≤ 10,000 international units (IU)/mL or unquantifiable or undetectable HCV RNA at screening
8. Previous use of an HCV direct-acting antiviral agent (DAA)
9. Consideration by the investigator, for any reason, that the participant was an unsuitable candidate to receive ABT-493, ABT-530, or RBV (RBV for cirrhotic subjects only)
10. For participants in Study Part 2 who were enrolling with compensated cirrhosis: past clinical evidence of Child-Pugh B or C Classification (score of > 6) or clinical history of liver decompensation, including ascites (noted on physical exam), bleeding varices, use of beta-blockers for portal hypertension or ascites, or hepatic encephalopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armen Asatryan, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gane E, Poordad F, Wang S, Asatryan A, Kwo PY, Lalezari J, Wyles DL, Hassanein T, Aguilar H, Maliakkal B, Liu R, Lin CW, Ng TI, Kort J, Mensa FJ. High Efficacy of ABT-493 and ABT-530 Treatment in Patients With HCV Genotype 1 or 3 Infection and Compensated Cirrhosis. Gastroenterology. 2016 Oct;151(4):651-659.e1. doi: 10.1053/j.gastro.2016.07.020. Epub 2016 Jul 25. PMID 27456384
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Naganuma A, Chayama K, Notsumata K, Gane E, Foster GR, Wyles D, Kwo P, Crown E, Bhagat A, Mensa FJ, Otani T, Larsen L, Burroughs M, Kumada H. Integrated analysis of 8-week glecaprevir/pibrentasvir in Japanese and overseas patients without cirrhosis and with hepatitis C virus genotype 1 or 2 infection. J Gastroenterol. 2019 Aug;54(8):752-761. doi: 10.1007/s00535-019-01569-7. Epub 2019 Mar 13. PMID 30868245
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- [Derived] Kwo PY, Poordad F, Asatryan A, Wang S, Wyles DL, Hassanein T, Felizarta F, Sulkowski MS, Gane E, Maliakkal B, Overcash JS, Gordon SC, Muir AJ, Aguilar H, Agarwal K, Dore GJ, Lin CW, Liu R, Lovell SS, Ng TI, Kort J, Mensa FJ. Glecaprevir and pibrentasvir yield high response rates in patients with HCV genotype 1-6 without cirrhosis. J Hepatol. 2017 Aug;67(2):263-271. doi: 10.1016/j.jhep.2017.03.039. Epub 2017 Apr 13. PMID 28412293

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population: all participants who received at least 1 dose of study drug. Two participants assigned to Arm I received the incorrect dose of study drug throughout their participation in the study (ABT-493 200 mg QD instead of 300 mg) and are therefore included in Arm A instead of Arm I in the safety population.
Period: Enrolled
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Started | 40 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 34 | 0 | 34
Completed | 40 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 34 | 0 | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treated
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Started | 42 (Two Arm I participants received ABT-493 doses of 200 mg instead of 300 mg and are included in Arm A) | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 32 (Two Arm I participants received ABT-493 doses of 200 mg instead of 300 mg and are included in Arm A) | 0 | 34
Completed Treatment | 42 | 38 | 0 | 0 | 0 | 27 | 0 | 0 | 32 | 0 | 33
Completed | 41 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 31 | 0 | 31
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study drug. Two participants assigned to Arm I received the incorrect dose of study drug throughout their participation in the study (ABT-493 200 mg QD instead of 300 mg) and are therefore included in Arm A instead of Arm I in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K | Total
Number analyzed (Participants) | 42 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 32 | 0 | 34 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.01) | 52.5 (10.41) |  |  |  | 58.9 (5.47) |  |  | 55.0 (11.13) |  | 53.5 (10.34) | 54.1 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 0 | 0 | 0 | 7 | 0 | 0 | 16 | 0 | 15 | 76
  Male | 25 | 18 | 0 | 0 | 0 | 20 | 0 | 0 | 16 | 0 | 19 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks Post-treatment
Description: The percentage of participants with sustained virologic response (plasma hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intention-to-treat population: all participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 40 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 34 | 0 | 34
percentage of participants | 100 [91.2 to 100] | 97.4 [86.8 to 99.5] |  |  |  | 96.3 [81.7 to 99.3] |  |  | 100 [89.8 to 100] |  | 97.1 [85.1 to 99.5]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 4 Weeks Post-treatment
Description: The percentage of participants with sustained virologic response (plasma hepatitis C virus ribonucleic acid [HCV RNA] less than the lower limit of quantification [<LLOQ]) 4 weeks after the last dose of study drug.
Time Frame: 4 weeks after the last actual dose of study drug
Population: Intention-to-treat population: all participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 40 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 34 | 0 | 34
percentage of participants | 100 [91.2 to 100] | 97.4 [86.8 to 99.5] |  |  |  | 96.3 [81.7 to 99.3] |  |  | 100 [89.8 to 100] |  | 100 [89.8 to 100]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: The percentage of participants with on-treatment virologic failure (defined as confirmed hepatitis C virus ribonucleic acid (HCV RNA) greater than or equal to the lower limit of quantitation [≥ LLOQ] after HCV RNA < LLOQ during treatment), confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Screening, Day 1, Day 3, treatment weeks 1, 2, 4, 6, 8, 10, and 12 or premature discontinuation from treatment
Population: Intention-to-treat population: all participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 40 | 39 | 0 | 0 | 0 | 27 | 0 | 0 | 34 | 0 | 34
percentage of participants | 0 [0.0 to 8.8] | 0 [0.0 to 9.0] |  |  |  | 0 [0.0 to 12.5] |  |  | 0 [0.0 to 10.2] |  | 0 [0.0 to 10.2]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed hepatitis C virus ribonucleic acid (HCV RNA) greater than or equal to the lower limit of quantitation (≥ LLOQ) between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K
Number analyzed (Participants) | 40 | 38 | 0 | 0 | 0 | 27 | 0 | 0 | 34 | 0 | 33
percentage of participants | 0 [0.0 to 8.8] | 2.6 [0.5 to 13.5] |  |  |  | 3.7 [0.7 to 18.3] |  |  | 0 [0.0 to 10.2] |  | 0 [0.0 to 10.4]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug, up to 16 weeks. Serious adverse events were collected starting after the study-specific informed consent was signed and continuing until 30 days after the last dose of study drug, up to 23 weeks.
Groups:
- Arm B: ABT-493 200 mg once daily (QD) + ABT-530 40 mg QD for 12 weeks in HCV genotype 1-infected participants without cirrhosis
- Arm F: ABT-493 200 mg once daily (QD) + ABT-530 120 mg QD for 12 weeks in HCV genotype 1-infected participants with compensated cirrhosis
- Arm I: ABT-493 300 mg once daily (QD) + ABT-530 120 mg QD for 12 weeks in HCV genotype 4-, 5-, and 6- infected participants without cirrhosis
- Arm K: ABT-493 300 mg once daily (QD) + ABT-530 120 mg QD for 8 weeks in HCV genotype 1-infected participants without cirrhosis
Arm/Group | Arm A | Arm B | Arm F | Arm I | Arm K
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/39 | 1/27 | 0/32 | 1/34
Other Adverse Events (participants affected / at risk) | 22/42 | 22/39 | 9/27 | 20/32 | 19/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=42) | Arm B (N=39) | Arm F (N=27) | Arm I (N=32) | Arm K (N=34)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=42) | Arm B (N=39) | Arm F (N=27) | Arm I (N=32) | Arm K (N=34)
VISION BLURRED (Eye disorders) | 0 | 1 | 0 | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 3 | 3 | 1 | 5 | 3
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
FLATULENCE (Gastrointestinal disorders) | 3 | 0 | 0 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 5 | 8 | 0 | 3 | 3
FATIGUE (General disorders) | 10 | 5 | 3 | 3 | 6
PAIN (General disorders) | 1 | 1 | 0 | 1 | 2
PYREXIA (General disorders) | 3 | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 2 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 3
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 2
DIZZINESS (Nervous system disorders) | 2 | 2 | 0 | 2 | 1
HEADACHE (Nervous system disorders) | 5 | 8 | 3 | 8 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 2 | 3 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 2 | 0 | 1 | 2 | 0
INSOMNIA (Psychiatric disorders) | 1 | 3 | 0 | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3
PARANASAL SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.